CLINICAL TRIAL: NCT04138238
Title: Post-market Registry to Evaluate the Safety and Efficacy of the Supraflex Cruz Sirolimus-eluting Coronary Stent System in the Treatment of All-comer Patients With Coronary Artery Disease
Brief Title: Cruz HBR Registry - Post-market Registry to Evaluate the Safety and Efficacy of the Supraflex Cruz Stent
Status: Completed | Type: Observational
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: SMT CT 2019-20/108
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
Keywords: Supraflex Cruz; Sirolimus-eluting Stent; High Bleeding Risk; Coronary Artery Disease; Arteriosclerosis; Myocardial Ischemia; Vascular Diseases; Coronary Intervention; Observational Registry; Ultra-thin Strut Biodegradable Polymer
MeSH Terms: conditions — Coronary Artery Disease; Arteriosclerosis; Myocardial Ischemia; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supraflex Cruz Sirolimus-eluting Stent
  Interventions: Device: Supraflex Cruz Sirolimus-eluting Stent

INTERVENTIONS:
Device: Supraflex Cruz Sirolimus-eluting Stent — Patient implanted with at least one Supraflex Cruz sirolimus-eluting stent as a part of planned clinical care

SUMMARY:
This is a prospective, multicenter, open-label, single-arm registry. The primary objective of this registry is to confirm the results of the Supraflex Cruz stent in real life all-comer patients (800 patients as in the Supraflex arm of the TALENT trial) and demonstrate that the Supraflex Cruz stent is not inferior to the BioFreedom stent in High Bleeding Risk (HBR) patients (400 patients) with respect to device oriented composite endpoint (DOCE) at 12 months. All patients will be followed up to 12 months after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. De novo or re-stenotic significant stenosis in at least one native coronary artery
3. Patients with silent ischemia, stable angina, unstable angina or non-STEMI eligible for PCI (no limitation of the number of treated lesions and vessels, except higher tercile of Syntax score assessed by the site)
4. Target lesions suitable for PCI with Drug-eluting Stent (DES) diameter between 2.00 and 4.50 mm
5. Total lesion length should be from 15 to 120 mm
6. Patient is willing and capable to sign the written informed consent and comply with all requirements of the registry
7. Planned staged procedures are allowed within 3 months using Supraflex Cruz stent only

Exclusion Criteria:

1. SYNTAX Score > 32
2. Hemodynamic instability or cardiogenic shock
3. Known hypersensitivity or contraindication to any component of the study stent or the eluting drug, to media contrast, to dual antiplatelet therapy (DAPT) medication required by current practice
4. Subject is pregnant, nursing or is a woman with child-bearing potential
5. Any co-morbid condition with life expectancy < 1 year or that may result in protocol non-compliance
6. Patients who are participating in another drug or device investigational study, which has not reached its primary endpoint
7. Patients under judicial protection, tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comer patients affected by silent ischemia, stable angina or acute coronary syndrome (unstable angina and non-STEMI), who qualify for percutaneous coronary intervention (PCI), 400 patients of the population must qualify for HBR criteria
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Device Oriented Composite Endpoint (DOCE) | 12 months
  DOCE is a composite of cardiovascular death, myocardial infarction (MI) not clearly attributable to a non-target vessel and clinically-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
All death, cardiovascular death and non-cardiovascular death | 6 months and 12 months
All myocardial infarction (MI) | 6 months and 12 months
Target vessel MI and MI not clearly attributable to non-target vessel | 6 months and 12 months
Clinically indicated target lesion revascularization (TLR) | 6 months and 12 months
All target lesion revascularization (TLR) | 6 months and 12 months
  Clinically and non-clinically indicated target lesion revascularization (TLR)
All target vessel revascularization (TVR) | 6 months and 12 months
  Clinically and non-clinically indicated target vessel revascularization (TVR)
All revascularization | 6 months and 12 months
  Any revascularization, TLR (clinically and non-clinically), TVR (clinically and non-clinically) and non-TVR
Stent thrombosis (ARC2) | 6 months and 12 months
Device success | Up to 1 Day
  Defined as deployment of the stents without system failure or device-related complication
Lesion success | Up to 1 Day
  Defined as the attainment of < 50% residual stenosis of the target lesions post-PCI
Procedure success | Up to 7 Days
  Defined as all lesion successfully treated without the occurrence of DOCE during the hospital stay
Major bleeding (BARC 3 to 5) in the HBR population | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Christoph K Naber, PD. Dr. Med., Principal Investigator — Klinikum Wilhelmshaven
Locations (26):
- France (6):
  - Centre Hospitalier Haguenau, Haguenau
  - Hôpital Privé Jacques Cartier, Massy
  - CHRU de Montpellier, Montpellier
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart
  - Clinique Saint Hilaire, Rouen
  - CHU de Toulouse - Rangueil, Toulouse
- Germany (17):
  - Kerckhoff Heart Center, Bad Nauheim
  - Heart and Diabetes Center Nordrhine Westfalia, Bad Oeynhausen
  - Segeberg Kliniken, Bad Segeberg
  - Charité Campus Mitte, Berlin
  - Charité Campus Benjamin Franklin, Berlin
  - Charité Campus Virchow, Berlin
  - St Johannes Hospital, Dortmund
  - Herzzentrum Dresden - Universitätklinikum an der TU Dresden, Dresden
  - Praxisklinik Dresden, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - University Hospital Erlangen, Erlangen
  - Elizabeth Krankenhaus, Essen
  - UKSH, Kiel
  - Universität Leipzig - Herzzentrum, Leipzig
  - Städtische Kliniken Neuss, Lukaskrankenhaus, Neuss
  - Universitätsklinikum, Regensburg
  - Klinikum Wilhelmshaven, Wilhelmshaven
- Switzerland (3):
  - University and Hospital Fribourg, Fribourg
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No